CLINICAL TRIAL: NCT03589820
Title: Clinical Efficacy of Artificial Liver Support System Using Combination of Plasma Exchange and Continuous Hemodiafiltration in Treatment of Wilson's Disease - Related Liver Failure
Brief Title: Plasma Exchange and Continuous Hemodiafiltration in Treatment of Wilson's Disease-related Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XWX1
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Wilson Disease; Liver Failure
Keywords: Wilson Disease; Liver Failure; plasma exchange; continuous hemodiafiltration
MeSH Terms: conditions — Hepatolenticular Degeneration; Liver Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial liver support system group (Active Comparator): 30 patients will receive treatment of artificial liver support system using combination of plasma exchange and continuous hemodiafiltration and internal medicine.
  Interventions: Other: artificial liver support system
- Control group (No Intervention): 30 patients will receive treatment of internal medicine.

INTERVENTIONS:
Other: artificial liver support system — Patients will receive the treatment of artificial liver support system using combination of plasma exchange and continuous hemodiafiltration and internal medicine. The volume of fresh frozen plasma used in plasma exchange is 2000 millilitre. The time for continuous hemodiafiltration is about 8 hours.
  Arms: Artificial liver support system group

SUMMARY:
This study is to investigate the clinical efficacy of artificial liver support system using combination of plasma exchange and continuous hemodiafiltration in treatment of Wilson's Disease - related liver failure. 30 patients will receive treatment of plasma exchange and continuous hemodiafiltration and internal medicine. 30 patients will receive treatment of internal medicine.

DETAILED DESCRIPTION:
Wilson's disease (WD) is an inherited disorder in which defective biliary excretion of copper leads to its accumulation, particularly in liver and brain. Presenting symptoms of liver disease can be highly variable, ranging from asymptomatic, with only biochemical abnormalities, to overt cirrhosis with all its complications. Acute liver failure (ALF) presentation is the most dramatic and may arise with catastrophic suddenness. It is considered rare, constituting only 3% of ALF cases in the pediatric ALF series in USA and associated with a high mortality reaching 95%. Patients with acute liver failure due to WD require liver transplantation, which is lifesaving. Kido J et al reported clinical outcomes of patients with liver failure were improved by artificial liver support system using combination of plasma exchange and continuous hemodiafiltration. So the investigators design this protocol: 30 patients will receive treatment of plasma exchange and continuous hemodiafiltration and internal medicine, 30 patients will receive treatment of internal medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Wilson Disease: serum ceruloplasmin < 0.2g/L, 24 hours urinary copper > 40μg, Kayser-Fleischer ring present;
2. Do not receive drugs to promote the excretion of copper ever before;
3. Serum total bilirubin > 10 times upper limit of normal, prothrombin time activity < 40% or prothrombin time international ratio > 1.5.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-28 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | 48 weeks
  Whether patients will survive is observed in the follow-up.

SECONDARY OUTCOMES:
liver function improvement | 48 weeks
  Symptoms (i.e. fatigue, appetite, nausea, vomiting, jaundice, consciousness) and laboratory tests (i.e. blood cells, alanine transaminase, total bilirubin, prothrombin time, creatinine, ceruloplasmin, serum copper) are observed in the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided